CLINICAL TRIAL: NCT02888561
Title: The Impact of Dobutamine and Nitrite on Myocardial Supply and Demand in Heart Failure
Brief Title: Haemodynamic Effects of Dobutamine and Nitrite in LV Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 199826
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Dobutamine; Nitrites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dobutamine — Dobutamine will be infused at the time of coronary angiography while coronary and LV haemodynamics are measured using a Combowire (dual pressure and flow sensor tip guide wire) and left ventricular conductance catheter.
Drug: Nitrite — Nitrite will be infused at the time of coronary angiography while coronary and LV haemodynamics are measured using a Combowire (dual pressure and flow sensor tip guide wire) and left ventricular conductance catheter.

SUMMARY:
Patients with poor heart function can, in certain situations, have a further weakening of the heart muscle such that it becomes difficult to provide enough blood to the brain and other organs. In these cases, heart function can be supported by the use of medicines or heart pumps. One of the most widely used medicines is Dobutamine, given as an infusion (a drip). Although Dobutamine has been in use for decades and does improve blood flow to the organs, previous studies have not shown any impact on recovery of heart muscle function and survival. Key to unravelling this discrepancy is to understand the precise effects of Dobutamine on the oxygen supply to, and oxygen usage by, the heart muscle. We also aim to find out whether simultaneous infusion of another drug called Nitrite (naturally occurring substance that is found in beetroot for example, much like GTN) can enhance the beneficial effects of Dobutamine on the oxygen supply-demand balance of the heart. In recent years, major advances in technology mean that it is now possible to obtain this information in patients undergoing coronary angiography procedures by making detailed measurements of heart muscle function and blood flow in the heart arteries using a conductance catheter (measures volume and pressure within the main pumping chamber of the heart) and the Combowire (dual pressure and flow sensor tip angioplasty guidewire). The aim of this study is to understand the effect of a brief infusion of Dobutamine and nitrite on heart muscle function, oxygen supply and oxygen usage through this use of this technology, directly following the patients routine coronary angiogram. Patients will have these measurements taken using the technology described above during the infusion of both dobutamine and nitrite, inserted through blood vessels that reach the heart.

ELIGIBILITY:
Inclusion Criteria:

1. Left Ventricular Ejection Fraction <40%
2. Patients aged >18 years
3. Able to provide written consent

Exclusion Criteria:

1. Known acquired or congenital structural heart disease such as severe valve disease, ventricular/atrial septal defects
2. Haemodynamic Instability
3. Severe disease in major proximal coronary arteries or planned percutaneous coronary intervention during the index procedure

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for diagnostic coronary angiography following a diagnosis of heart failure, with a left ventricular ejection fraction of less than or equal to 40%.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Coronary Flow (average peak velocity) | During procedure.
left ventricular stroke work | during procedure

SECONDARY OUTCOMES:
rate pressure product | during procedure
pressure volume area | during procedure
coronary microvascular resistance | during procedure
stroke volume | during procedure
Distal tissue perfusion | during procedure
Magnitude of forward compression wave | during procedure
magnitude of backward expansion wave | during procedure

CONTACTS AND LOCATIONS:
Locations (1):
- British Heart Foundation Centre of Excellence, The Rayne Institute, KCL, at Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No